CLINICAL TRIAL: NCT00035958
Title: Toward Improved Understanding of Pathogenesis and Treatment of Childhood Onset Dermatomyositis
Brief Title: Understanding the Pathogenesis and Treatment of Childhood Onset Dermatomyositis
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Incorporating the recommendations of the NIH-formed DSMB in the study procedures would make the project budget over the limit for this funding mechanism.
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); Immunex Corporation (Industry)
Responsible Party: Daniel J. Lovell, MD, MPH, Cincinnati Children's Hospital Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P60AR047784 (NIH); P60AR047784 (NIH); NIAMS-078
Record Dates: First submitted 2002-05-07; First posted 2002-05-08 (Estimated); Last update posted 2013-08-01 (Estimated); Status verified 2013-07

CONDITIONS: Dermatomyositis
Keywords: Juvenile Dermatomyositis; Pediatric; Randomized Clinical Trial; Pediatric Rheumatology
MeSH Terms: conditions — Dermatomyositis | interventions — Prednisone; Methotrexate; Etanercept

INTERVENTIONS:
Drug: Prednisone
Drug: Methotrexate
Drug: Etanercept

SUMMARY:
Juvenile dermatomyositis (JDMS) is one of the most serious of the childhood rheumatic diseases. The theory behind this trial is that early introduction of etanercept or methotrexate will prove to be effective in the treatment of JDMS. Pretreatment muscle biopsies, we believe there will be abnormalities in the blood vessels that will be correlated with worse physical strength and daily functional ability. The long-term goal is to improve the treatment of this serious childhood onset rheumatic disease and to better understand the pathogenic mechanism for the development of the vasculopathy (disorder of blood vessels) of JDMS. Identification of the specific mechanism of the vasculopathy may allow for the rational introduction of biologic treatments focused on vascular growth.

DETAILED DESCRIPTION:
The mortality of JDMS is 3-39% with over 40% of patients demonstrating long-term disability. Current first line therapy is high-dose corticosteroids with the attendant significant drug-related toxicity. Over 30% of JDMS patients fail to respond adequately to steroids and require additional immunosuppression, none of which have been tested in prospective, randomized, controlled trials. The unique occlusive vasculopathy in JDMS is critical in the pathogenesis and predictive of prognosis but poorly understood. Elevated levels of tumor necrosis factor (TNF) alpha have been shown to be present in JDMS and are associated with a more severe and chronic course.

Seventy-five children with definite JDMS will be enrolled in a 24-month prospective, randomized, multicentered trial comparing 3 treatments: oral prednisone (P), combination of oral prednisone and methotrexate (P/MTX), and combination of oral prednisone and etanercept (P/E). Primary response measures will be muscle strength and mean duration of steroid therapy. Secondary response variables are disability in daily function and height and weight growth velocity (steroid toxicity measures). The combination of P/E will be tested and compared to both P alone and the combination of P/MTX after 3, 6, 12, 18, and 24 months of treatment. In addition, the combination of P/MTX will be compared to P alone after 3, 6, 12, 18, and 24 months of treatment. In pretreatment muscle biopsies, proangiogenic factors (such as vascular endothelial cell growth factor and basic fibroblast growth factor), angiostatic factors (such as angiostatin and endostatin), and vascular morphology (vessel number, width, length and area) will be quantified and tested for ability to predict muscle strength and functional ability 3, 6, 12, 18, and 24 months later.

ELIGIBILITY:
Inclusion criteria at the time of enrollment:

* Definite or probable diagnosis of JDMS by the criteria of Bohan and Peter
* No prior systemic steroid treatment for JDMS
* If able to become pregnant (females) or impregnate (males) and are sexually active, then must have negative serum pregnancy test at baseline and be utilizing effective form of birth control
* Patient and/or parent or legal guardian must be willing to sign consent and assent forms

Exclusion criteria at the time of enrollment:

* History of chronic or recurrent infections sufficient to preclude the use of etanercept
* Prior treatment with specific TNF-blocking agents
* Demonstration of cutaneous or gastrointestinal (GI) ulceration at the time of diagnosis
* JDMS-related pulmonary disease at time of diagnosis (interstitial lung disease or aspiration pneumonia confirmed by radiograph)
* JDMS-related cardiomyopathy (echocardiogram confirmation)
* Any uncontrolled, clinically significant pre-existent systemic disease (hepatic, renal, neurological, endocrine, cardiac, gastrointestinal, or hematologic disease) within 24 weeks of start of study
* Known HIV, hepatitis B surface antigen not related to vaccination, or hepatitis C antibody positivity
* Pregnant or nursing female
* Any of the following laboratory abnormalities at baseline: platelet count < 100,000/cmm, total white cell count of < 3000 cells/cmm, neutrophils < 1000 cells/cmm, serum bilirubin > 2 times upper limit of normal, estimated creatinine clearance of < 90 mL/min/1.73 M2 BSA estimated by formula for males age 2 to <13 (0.55 X ht in cms/serum creatinine), age 13-18 (0.7 X ht in cms/serum creatinine) and females age 2-18 (0.55 X ht in cms/serum creatinine)
* Received live virus vaccination within 3 months prior to study entry (contraindication for MTX or etanercept therapy)
* Past or current substance abuse or psychiatric history that would interfere with ability to give informed consent or comply with study requirements or physician instructions

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75
Dates: Start 2002-08; Primary Completion 2002-08 (Actual); Study Completion 2002-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J. Lovell, MD, MPH, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio, United States